CLINICAL TRIAL: NCT07187596
Title: Progressive Elaboration Framework of Mortality in Treated and Controlled Hypertension: A Pooled Analysis of Contributing Factors to Silent or Uncontrollable Fatal Syndromes
Brief Title: Mortality Outcome of Controlled Hypertension
Acronym: MOCH
Status: Recruiting | Type: Observational
Sponsor: DejthidaNathaphong (Other)
Responsible Party: Principal Investigator, Nathaphong Dejthida, Principle Investigator, DejthidaNathaphong
Other Study IDs: NathaphongDejthida
Record Dates: First submitted 2025-09-09; First posted 2025-09-23 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Hypertension; Morality; Death; Pre-Eclampsia; Cardiovascular Diseases; Stroke; Renal Disease; Artery Stenosis; Arterial Aneurysm; Arterial Rupture; Maternal Death
Keywords: Controlled blood pressure; Mortality outcomes
MeSH Terms: conditions — Hypertension; Death; Pre-Eclampsia; Cardiovascular Diseases; Stroke; Kidney Diseases; Maternal Death

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This pooled analysis investigates death outcomes in patients with pharmacologically treated and blood pressure-controlled hypertension. Despite documented BP control, some patients still suffer fatal cardiovascular, cerebrovascular, renal, or unexplained syndromes. This study aims to synthesize available evidence across study types to identify treatment pitfalls, contributing syndromes, and non-BP factors associated with these fatal outcomes.

DETAILED DESCRIPTION:
Although hypertension is commonly treated and controlled to target levels, fatalities still occur in some patient subgroups. This pooled review seeks to identify and analyze these populations' contributing factors, comorbidities, treatment contexts, and physiological mechanisms associated with mortality. Data will be collected from peer-reviewed studies and registries. Statistical analysis will include descriptive synthesis, subgroup tabulations, and exploratory regression.

Open-label analysis aims to investigate death outcomes among patients with treated and well-controlled hypertension by synthesizing results from published clinical trials, observational studies, and systematic reviews.

The study will statistically evaluate endpoint include fatal cardiovascular, cerebrovascular, renal, or vascular events in patients in any arm with documented blood pressure control, with clearly seen evidence.

ELIGIBILITY:
Inclusion criteria

* Human studies (RCTs, cohort, case-control, registry studies, etc.) declare participants with treated and controlled hypertension manage (regardless of drug class, duration, or comorbidity) reported mortality outcomes: all-vascular death, cardiovascular death, sudden death, etc.
* Studies in any setting (outpatient, inpatient, long-term follow-up)
* Articles in English
* Full-text available

Exclusion criteria

* Animal specimen or parameter studies
* Uncontrolled studies (e.g., case series without control, phase I safety trials)
* No mortality endpoint reported
* Purely mechanistic studies or trials that do not address BP or survival directly
* Pediatric studies unless separated subgroup for treated hypertension is available
* Glaucoma or portal hypertension or Pulmonary Hypertension without essential/systemic hypertension outcomes
* Infection without direct declare that septic shock or immunological failure associated by vascular cause from systemic hypertension
* Secondary/post-hoc analyses that do not report original mortality data

Ages: 1 Minute to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Studies including patients (any age or sex) with:
  * Interventional treatment for hypertension
  * Documented blood pressure control (as defined by each primary study)
  * Reported mortality or fatal outcome
Sampling Method: Non-Probability Sample
Enrollment: 1000000 (Estimated)
Dates: Start 2025-09-18 (Actual); Primary Completion 2026-05-18 (Estimated); Study Completion 2026-07-14 (Estimated)

PRIMARY OUTCOMES:
All-cause vascular mortality | Day one until last follow up at least 24 hour to study completion date at least 30 days outcomes but not over 10 years
  Cardiovascular mortality (Cardiac-related death in controlled hypertension patients), cerebrovascular death(Stroke-related fatal outcomes in BP-controlled patients), renal occlusion/rupture/failure causing death (Mortality from renal failure in treated, controlled hypertensives), life-threatening vascular rupture, Major Adverse Cardiovascular Death or

SECONDARY OUTCOMES:
Sudden death | Day one until last follow up at least 24 hour to study completion date at least 30 days outcomes but not over 10 years
  Death suddenly with autopsy or complete CPR during collapse of cardiac or respiratory or brain arrested
End-organ failure leading to death | 90 days outcomes after participant recruitment (death/alive)
  Vascular abnormality causing failure of organ leading death with evidence by imaging, laboratory investigation or autopsy
ICU death | 90 days outcomes start with day 1 admit at ICU (death/alive)
  Systemic arterial hypertension is the main reason for admission at critical care unit report death
Maternal associated hypertension death | During pregnancy period from GA 1 week to delivery (pre-term, term-post-term) to 6 week follow up postpartum
  Mortality outcomes of hypertension during pregnancy both from gynecologic organ failure or systemic organ failure
Hypertension associated death in the young | Day one until last follow up at least 24 hour to study completion date at least 30 days outcomes but not over 18 years of ages of participant
  Mortality outcomes that clear defined high blood pressure of that age and declared mortality cause during or after any type of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nathaphong Dejthida, MD, Principal Investigator — DejthidaNathaphong
Locations (1):
- Owned study, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
The study already registered from PROSPERO number CRD420251072526
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: TIMELINE OF THE REVIEW Date of first submission to PROSPERO 01 July 2025 Review timeline Start date: 14 June 2025. End date: 31 December 2025.
  Date of registration in PROSPERO
  01 July 2025
Access Criteria: Public registered
URL: https://www.crd.york.ac.uk/PROSPERO/view/CRD420251072526

REFERENCES:
- See also: PROSPERO registry — https://www.crd.york.ac.uk/PROSPERO/view/CRD420251072526

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-25): https://cdn.clinicaltrials.gov/large-docs/96/NCT07187596/Prot_SAP_001.pdf